CLINICAL TRIAL: NCT00342706
Title: Building Healthy Teen Relationships and Reproductive Practices to Increase Interpregnancy Intervals
Brief Title: Building Healthy Teen Relationships and Reproductive Practices to Increase Intervals Between Pregnancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905083; 05-CH-N083
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-29

CONDITIONS: Teen Pregnancy
Keywords: Teen Pregnancy; Short Inter-Pregnancy Intervals

INTERVENTIONS:
Procedure: Community based intervention

SUMMARY:
This study will determine the best ways to help teen mothers stay healthy and to increase the time between their pregnancies to at least 2 years. It is designed to encourage attitudes and behaviors that are generally thought to be related to longer intervals between pregnancies. Children of teen mothers generally receive less health care, have lower IQ scores and are more likely to enter foster care. They have less supportive home environments and higher rates of incarceration and teen childbearing.

African-American and Latino teenagers living in the Washington, D.C., metropolitan area who are pregnant with their first baby may be eligible for this study. Mothers or mother figures of the teens also are encouraged to participate. Candidates must be between 15 and 18 year of age and speak English.

Teen mothers enrolled in the study take a urine pregnancy test every 6 months during this 2-year study. They are randomly assigned to one of the following two groups:

Usual Care Group: Teens in this group are interviewed by telephone for about 1 hour every 6 months and for about 15 minutes at 3, 9, 15 and 21 months. The hour-long interview includes questions about the teen's feelings and behaviors, risks to her health and well being, and how she communicates with her boyfriend and family members. She is also asked about what she does to reach personal goals, what she thinks about sexual health, and what support she gets from her family, boyfriend, or others. The 15-minute interview is an update to check on the teen's health and pregnancy status and to verify contact information.

Intervention Group: Teens in this group are asked the same questions as those in the usual care group; however, they are involved in a project designed to encourage them to set goals of furthering their education and training and wait at least 2 years before becoming pregnant again. Teens in this group are counseled on learning to communicate and work out problems with their family and boyfriend and on how to keep from getting pregnant again soon. The participants meet for a 2-hour group session every 3 months at a local health center and are contacted frequently by a cell phone, which is provided to them at no cost. The phone sessions are about things that are important to the teens, such as problems in their relationships, health, sexually transmitted diseases, and preventing another pregnancy too soon. The conversations are private and take about 45 minutes.

Mothers (or...

DETAILED DESCRIPTION:
The major objective of this program is to test the effectiveness of a community based intervention for minority teen mothers. The primary aim of the project is to: Evaluate the effectiveness of a community based intervention for minority teen mothers, with the primary purpose of increasing the inter-pregnancy interval to greater than 24 months. The secondary aim is to evaluate the effectiveness of a community based intervention for minority teen mothers, with a secondary purpose of improving knowledge, attitudes, behaviors, relationships and connectedness generally understood to be related to length of inter-pregnancy intervals.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following criteria will determine eligibility for the study:

1. African American and Latino primiparous pregnant or newly parenting (0-6 weeks);
2. Age 15-18 years inclusive; and
3. Teens who are 19 years old if they have not graduated from high school.

EXCLUSION CRITERIA:

1. Non-English speaking;
2. Any serious medical condition or disability that would interfere with the participant responding adequately to evaluation measures;
3. Obvious cognitive impairment that interferes in participating in informed consent;
4. Incarceration at enrollment or during the study.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 750 (Estimated)
Dates: Start 2005-01-10; Primary Completion 2011-04-29 (Actual); Study Completion 2011-04-29 (Actual)

PRIMARY OUTCOMES:
Delay of a subsequent pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aarons SJ, Jenkins RR, Raine TR, El-Khorazaty MN, Woodward KM, Williams RL, Clark MC, Wingrove BK. Postponing sexual intercourse among urban junior high school students-a randomized controlled evaluation. J Adolesc Health. 2000 Oct;27(4):236-47. doi: 10.1016/s1054-139x(00)00102-6. PMID 11008086
- [Background] Akinbami LJ, Cheng TL, Kornfeld D. A review of teen-tot programs: comprehensive clinical care for young parents and their children. Adolescence. 2001 Summer;36(142):381-93. PMID 11572313
- [Background] Blake SM, Ledsky R, Goodenow C, Sawyer R, Lohrmann D, Windsor R. Condom availability programs in Massachusetts high schools: relationships with condom use and sexual behavior. Am J Public Health. 2003 Jun;93(6):955-62. doi: 10.2105/ajph.93.6.955. PMID 12773362